CLINICAL TRIAL: NCT04882553
Title: The Relation Between Oesophageal Pressure and Diaphragm Thickening Fraction in Spontaneously Breathing Sedated Children: a Feasibility Study.
Brief Title: Pediatric Diaphragm Thickness Trial
Acronym: PeDia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, Tom Schepens, MD, data manager, University Hospital, Antwerp
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 21/15/208; 1653 (Other: EDGE); 21/15/208 (Other: IRB)
Record Dates: First submitted 2021-05-06; First posted 2021-05-12 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2021-09

CONDITIONS: Child
Keywords: diaphragm thickening fraction; oesophageal pressure

STUDY DESIGN:
Intervention Model Description: a single-centre physiological cohort study to evaluate the feasibility of using the thickening fraction as a parameter for diaphragm activity during spontaneous breathing in sedated children.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Incremental inspiratory effort (Experimental): Every participant will be subjected to a stepwise incremental inspiratory effort:
  1. Ventilated
  2. Baseline spontaneous breathing with deep anesthesia (minimal alveolar concentration 1.5)
  3. Spontaneous breathing with PEEP 10 and deep anesthesia (minimal alveolar concentration 1.5)
  4. Spontaneous breathing with PEEP 0 and deep anesthesia (minimal alveolar concentration 1.5)
  5. Spontaneous breathing with PEEP 0 and moderate anesthesia (minimal alveolar concentration 1.0)
  6. Spontaneous breathing with PEEP 0 and moderate anesthesia (minimal alveolar concentration 1.0) and added inspiratory threshold of +7cmH2O
  7. Spontaneous breathing with PEEP 0 and moderate anesthesia (minimal alveolar concentration 1.0) and added inspiratory threshold of +15cmH2O
  Interventions: Procedure: Diaphragmatic echography; Procedure: Measurement of esophageal pressure; Diagnostic Test: Registration of respiratory mechanics

INTERVENTIONS:
Procedure: Diaphragmatic echography — Echography of the diaphragm at the zone of apposition. End-inspiratory and/or end-expiratory thickness of the diaphragm will be measured in M-mode.
Procedure: Measurement of esophageal pressure — Pressure will be measured in the lower third of the esophagus using an esophageal balloon and pressure transducer.
Diagnostic Test: Registration of respiratory mechanics — Pressures and volumes will be registered by the Fluxmed respiratory monitor (MBMED, Argentina)

SUMMARY:
The evaluation of diaphragm function in ventilated patients is not easy. One option is to use esophageal pressure (Pes) measurements but recently, diaphragmatic ultrasound has proven itself as a useful tool in this setting. In adults the thickening fraction (TF), which describes the difference in thickness between end-inspiration and end-expiration, correlates with the diaphragmatic pressure-time product per breath (PTPdi), an esophageal pressure-derived work of breathing parameter. There is a lack of data that tells us whether the same is true in children. This physiological study intends to look at the correlation between esophageal pressures and thickening fraction assessed by ultrasound in a pediatric cohort of patients.

DETAILED DESCRIPTION:
The gold standard in evaluating lung mechanics is the esophageal pressure. And although diaphragm ultrasound has been reported to be feasible in assessing diaphragm activity in sedated patients, no study has thus far looked at the relationship between the ultrasound parameters (i.e. thickening fraction) and the esophageal pressure. This is a single-centre physiological cohort study to evaluate the feasibility of using the thickening fraction as a parameter for diaphragm activity during spontaneous breathing in sedated children. Data will be collected during an elective surgical procedure with a patient under general anesthesia. If the patient's legal representative provides written informed consent, the patient is enrolled in the study before start of the anesthetic procedure and the trial ends on the moment of removal of the laryngeal mask.The registration of the physiological data will not interfere with the surgery.The thickening fraction (using ultrasound) and pressure measurements will be performed simultaneously and repetitive during different loads on the respiratory system.Esophageal pressures (Pes) will be measured with a single air-filled balloon catheter(AVEA™ smarthcath pediatric 7 Fr, Vyaire Medical Inc., IL, USA). The balloon catheter will be inserted nasally after the induction of anesthesia. The catheter will then be connected to a pressure transducer (FluxMed, MBMED, Argentina). The appropriate placement will be checked by commonly used methods. Firstly, the appropriate depth of insertion will be estimated by measuring the nose-ear-xyphoid distance, which is the distance from the nose to the diaphragm. Secondly, the balloon catheter will be inserted more deeply than this predicted distance, placing it in the stomach, and a positive pressure swing when mild abdominal pressure is exerted on a slightly inflated balloon will be noted. Thirdly, when retracted into the esophagus, cardiac reflections on the pressure monitor will appear. Fourth, when applying positive pressure ventilation, we will look for a positive deflection on the pressure curve. The output from the pressure transducer will be saved from the Fluxmed respiratory mechanics monitor. Pes will be measured over at least five consecutive breaths selected at the end of the pressure recordings. Ultrasound recordings will be done with the BK 3500 ultrasound machine, using a linear high-resolution probe. The parameter measured is the distance between the pleura and peritoneum as seen on a 2D image. The thickness using B-mode ultrasound imaging at end expiration on 10cm H2O of positive end-expiratory pressure (PEEP) and on zero PEEP (ZEEP) will be assessed. Furthermore, the thickness with Mmode imaging, both at end-inspiration (TEI) and end-expiration (TEE) will be measured. A transducer will be placed on the right side of the body in the midaxillary line at the level of the 8th and 9th intercostal space, the so-called zone of apposition. The probe will be positioned perpendicular to the skin, and temporary markings will be applied to the skin. Subjects are positioned in a supine position. TEE will be measured just before the thickening start and TEI measured at maximal thickening. Measurements will be averaged out of three or more consecutive breaths. The thickening fraction (TF) is calculated as (TEI - TEE)/TEE and expressed as a percentage. Digital images will be stored and re-interpreted by a separate, blinded interpreter.The thickening fraction recordings will be repeated during different loads on the respiratory system, with varying the depth of anesthesia (mean alveolar concentration of anesthetic vapor - MAC) and different added respiratory loads with a threshold valve and different levels of PEEP. An anesthesia circle circuit with standard pediatric tubing will consistently be used. The lowest dose of opioids will be used to the extent clinically possible.

Condition #1: during positive pressure ventilation, no spontaneous breaths Condition #2: spontaneous, MAC 1.5, PEEP, no added respiratory load Condition #3: spontaneous, MAC 1.5, PEEP 10, no added respiratory load (only Tdi, no TF) Condition #4: spontaneous, MAC 1.5, ZEEP, no extra added respiratory load Condition #5: spontaneous, MAC 1, ZEEP, no added respiratory load Condition #6: spontaneous, MAC 1, ZEEP, 7 cm H2O added respiratory load Condition #7: spontaneous, MAC 1, ZEEP, 15 cm H2O added respiratory load

These different conditions will alter the work of breathing the diaphragm has to perform and will allow us to better correlate thickening fraction with esophageal pressure.Preceding this study, a reproducibility study will assess intra-observer reproducibility for the researcher doing the ultrasound measurements.

A power analysis is not possible, as this is the first study comparing these parameters in children. Data will be analyzed using the SPSS statistical software package (SPSS Inc., IL, USA). Continuous variables will be reported as median (interquartile range). Friedman test and Wilcoxon paired tests (with post hoc Bonferonni correction) will be used to assess differences between related variables. Correlations between TF and Pes will be calculated using the Spearman method and performed for the entire data set (including all four respiratory conditions of each patient) because of the limited sample size. Two-tailed p values less than 0.05 will be considered significant.

All precautions will be taken to prevent complications due to placement of the balloon catheter but nevertheless all adverse events will be assessed.

ELIGIBILITY:
Inclusion Criteria: The patient must be scheduled for elective surgery where spontaneous breathing and physical access to the chest during surgery are feasible

* The patient must require general anaesthesia
* The parents are able to give informed consent for inclusion in the study

Exclusion Criteria:

* The patient is mechanically ventilated before start of the study.
* The patient is not anticipated to breathe spontaneously for a substantial amount of time prior to emergence from anesthesia
* The patient is known or suspected to have an anatomical malformation or surgical correction of the diaphragm.
* The patient suffers from a disease that may impair diaphragmatic function:

  * Central neural disease at the level of the brain (Stroke, Arnold-Chiari malformation) and spinal cord (quadriplegia, spinal muscular atrophy, syringomyelia).
  * Neural disease of the phrenic nerve (Guillain-Barré syndrome, tumor compression).
  * Disorders of the neuromuscular junction.
  * Muscular diseases (muscular dystrophies, myositis (infectious, inflammatory, metabolic).

Ages: 28 Days to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2021-06-11 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Esophageal pressure (cmH2O) at increasing levels of respiratory effort in spontaneously breathing, sedated children. | Perioperatively
  Esophageal pressures are measured in the lower third of the esophagus using an esophageal balloon and registered by an external pressure transducer.
Diaphragmatic thickening fraction (%) at increasing levels of respiratory effort in spontaneously breathing, sedated children. | Perioperatively
  The diaphragmatic thickening fraction (%) is calculated as [thickness at end-inspiration (mm) - thickness at end-expiration (mm)] / thickness at end-expiration (mm) x 100%.
  Diaphragmatic thickness is measured by ultrasound.
Feasibility (% success) of measuring diaphragmatic thickening fraction in spontaneously breathing ventilated children | Perioperatively
  The rate of success of diaphragmatic ultrasound in children, calculated as count of successful measurements / [count of successful measurements + count of unsuccessful measurements] x 100%

SECONDARY OUTCOMES:
Diaphragm thickness (mm) at different levels of positive end-expiratory pressure in spontaneously breathing, sedated children. | Perioperatively
  Diaphragmatic thickness is measured by ultrasound.

CONTACTS AND LOCATIONS:
Overall Officials: Tom Schepens, MD, Principal Investigator — University Hospital, Antwerp
Locations (1):
- University Hospital Antwerp, Edegem, Antwerp, Belgium

REFERENCES:
- [Derived] De Meyer GR, Flamey L, Adriaensens I, Van der Aerschot M, Van de Walle H, Vanmarsenille I, Jorens PG, Goligher EC, Saldien V, Schepens T. The Relationship Between Esophageal Pressure and Diaphragm Thickening Fraction in Spontaneously Breathing Sedated Children: A Feasibility Study. Pediatr Crit Care Med. 2023 Aug 1;24(8):652-661. doi: 10.1097/PCC.0000000000003248. Epub 2023 Apr 24. PMID 37092829